CLINICAL TRIAL: NCT04866355
Title: Short-term Effects of Lumbar Spine Manipulation Versus Pharmacological Therapy in Young Women With Primary Dysmenorrhea: a Randomized Controlled Trial.
Brief Title: Lumbar Spine Manipulation Versus Pharmacological Therapy in Young Women With Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Prof. Dr. Daniel Pecos Martín, Doctor, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2111730
Record Dates: First submitted 2021-04-23; First posted 2021-04-29 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Women With Primary Dysmenorrhea
MeSH Terms: interventions — Scopolamine; Ibuprofen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lumbar spine manipulation (Experimental): Application of lumbar spine manipulation by a physical therapist.
  Interventions: Other: Lumbar spine manipulation
- Lumbar spine manipulation plus pharmacological therapy (Active Comparator): Application of lumbar spine manipulation by a physical therapist along with pharmacological therapy.
  Interventions: Other: Lumbar spine manipulation; Drug: Hyoscine and Ibuprofen
- Pharmacological therapy (Active Comparator): Application of pharmacological therapy
  Interventions: Drug: Hyoscine and Ibuprofen

INTERVENTIONS:
Other: Lumbar spine manipulation — Lumbar spine manipulation
  Arms: Lumbar spine manipulation; Lumbar spine manipulation plus pharmacological therapy
Drug: Hyoscine and Ibuprofen — hyoscine (20 mg) and ibuprofen (400 mg) administered by oral via.
  Arms: Lumbar spine manipulation plus pharmacological therapy; Pharmacological therapy

SUMMARY:
Many treatments like acupuncture, manipulative therapy and pharmacological therapy have been proposed to alleviate symptoms associated with dysmenorrhea. However, no study has previously compared lumbar spine manipulation to pharmacological therapy in the treatment of primary dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* Presented with persistent primary dysmenorrhea lasting for three or more consecutive menstrual periods
* Presented menstrual cycles no longer than 35 days

Exclusion Criteria:

* Presented any other gynecological pathologies
* Systemic diseases
* Previous surgical interventions for gynecological complaints
* Depression
* Were receiving any other treatment for primary dysmenorrhea.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-02-28 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Change from baseline at 3 days
  Pain intensity measured with a visual analogue scale

SECONDARY OUTCOMES:
Pressure pain threshold measured in tibialis malleolus | Change from baseline at 3 days
  Pressure pain threshold measured with an algometer in tibialis malleolus
Pressure pain threshold measured in peroneal malleolus | Change from baseline at 3 days
  Pressure pain threshold measured with an algometer in peroneal malleolus
Low-back related disability | Change from baseline at 1 month
  Low-back related disability measured with the Oswestry Disability Index
Anxiety and depression | Change from baseline at 1 month
  Anxiety and depression measured with the Hospital Anxiety and Depression Scale

CONTACTS AND LOCATIONS:
Locations (2):
- Adelina Jazmin Castillo-Sanchez, Puebla City, Mexico
- Ruben Fernandez-Matias, Alcalá de Henares, Spain